CLINICAL TRIAL: NCT01275872
Title: A Randomized Clinical Trial on the Effect of Guided Imagery and Progressive Muscle Relaxation for the Management of Pain, Stress, Anxiety and Depression as a Means to Improve the Psychological Well-being and the Quality of Life for Patients With Breast and Prostate Cancer
Brief Title: Effect of Guided Imagery and Progressive Muscle Relaxation as a Means to Improve the Psychological Well-being and the Quality of Life for Patients With Breast and Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Lecturer-Researcher, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AC-GIPMR-85
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: guided imagery; progressive muscle relaxation; complimentary and alternative medicine; quality of life; stress; pain; anxiety
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Pain; Anxiety Disorders | interventions — Imagery, Psychotherapy; Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Guided Imagery and Progressive Muscle Relaxation (Experimental)
  Interventions: Other: Guided Imagery and Progressive Muscle Relaxation

INTERVENTIONS:
Other: Guided Imagery and Progressive Muscle Relaxation — 4 supervised sessions per patient for 4 weeks additional to daily unsupervised sessions

SUMMARY:
The purpose of this study is to determine whether Guided Imagery and Progressive Muscle Relaxation techniques are effective in the management of pain, fatigue, nausea-vomit, anxiety and depression in patients with either prostate or breast cancer.

This study includes a total of 200 patients with prostate and breast cancer randomly assigned to either a control or intervention group.

The intervention group received in total 4 sessions of Guided Imagery (protocol floating on a cloud) and Progressive Muscle Relaxation (breathing exercises and use of 11 groups of muscle progressively tensing and relaxing).

Measurements included the assessment of pain, fatigue, nausea-vomit, depression, anxiety and quality of life. Additionally, saliva samples were collected prior and after the sessions as to assess saliva cortisol and saliva α-amylase.

The same measurements were received by the patients of the control group as to allow comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast or prostate cancer
* Must be able to follow instructions
* Good cognitive ability
* Willing to participate

Exclusion Criteria:

* Use of cortisone
* Xerostomia
* oral mucositis

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Stress | 20 months
  Saliva α-amylase and saliva cortisol

SECONDARY OUTCOMES:
Quality of Life | 20 months
Fatigue | 20 months
Anxiety | 20 months
Depression | 20 months
Nausea-vomit | 20 months
Pain | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas I Charalambous, PhD, Principal Investigator — Cyprus University of Technology
Locations (1):
- Bank of Cyprus Oncology Centre, Nicosia, Nicosia, Cyprus

REFERENCES:
- [Derived] Charalambous A, Giannakopoulou M, Bozas E, Paikousis L. Parallel and serial mediation analysis between pain, anxiety, depression, fatigue and nausea, vomiting and retching within a randomised controlled trial in patients with breast and prostate cancer. BMJ Open. 2019 Jan 24;9(1):e026809. doi: 10.1136/bmjopen-2018-026809. PMID 30679301
- [Derived] Charalambous A, Giannakopoulou M, Bozas E, Marcou Y, Kitsios P, Paikousis L. Guided Imagery And Progressive Muscle Relaxation as a Cluster of Symptoms Management Intervention in Patients Receiving Chemotherapy: A Randomized Control Trial. PLoS One. 2016 Jun 24;11(6):e0156911. doi: 10.1371/journal.pone.0156911. eCollection 2016. PMID 27341675